CLINICAL TRIAL: NCT00159601
Title: Quality of Life and Mental Health in Children and Adolescents in a Child and Adolescent Psychiatric Outpatient Clinic and in the Normal Population
Brief Title: Quality of Life and Mental Health in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Council for Mental Health (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: NTNU-47019800
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Psychiatric Diagnosis; Mental Disorders
Keywords: Quality of Life; Mental health; Children; Adolescents; Normal population
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- outpatients in Child and Adolescent Mental Health Service
- youth from general population

SUMMARY:
The purpose of this study is to investigate different aspects of Quality of Life and mental health in patients under treatment in a child and adolescent psychiatric outpatient clinic and in the normal population.

DETAILED DESCRIPTION:
Measuring and monitoring Quality of Life in children and youths continues to increase in importance to both researchers and decision makers. Only a limited number of well validated instruments that measure Quality of Life in children exists, and in Norway only few has been translated into Norwegian. Up to date there are no studies investigating the quality of Life in Norwegian child and adolescent psychiatric patients in a longitudinal perspective, compared to the normal population.

Two generic Quality of Life instruments (KINDL, Bullinger & Ravens-Sieberer 2000 and the ILC, Matejatt & Remschmidt 1998) are introduced in Norway by this study in addition to the use of other well established measures like the "Child behaviour Check List" (Achenbach et al. 2001), etc.

Comparisons: 400 patients and their parents in a child psychiatric outpatient clinic 2000 pupils from the normal population in the middle of Norway Repeated measures after 6 months in both groups. In addition a follow up study for the clinical group 3 years after referral started in june 2006.

ELIGIBILITY:
Inclusion Criteria:

* All children 9-16 years of age, attending the 4th, 6th, 8th or 10th grades at public or private schools with at least 50 pupils, in the period from the 1st of September 2004 until 15th of July 2005 in the county of Sør-Trøndelag. Subjects and parents have to give their informed consent.
* All patients 8-10 years of age consecutively referred to to the child psychiatric outpatient clinic in the period from the 1st of June 2003 until 31st of December 2005, having a minimum of two direct contacts with the clinical staff. Patients and parents have to give their informed consent.
* Follow up: Three years after the patients met at the outpatient clinic for the first time.

Exclusion Criteria:

* Pupils lacking sufficient competence in the Norwegian language, due to foreign background or having a mental developmental level of more than two grades under the respective grade.
* Patients with psychosis or serious mental retardation.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients 8-10 years of age consecutively referred to the child psychiatric outpatient clinic in the period from 1th of June 2003 until 31th of December 2005, having a minimum of two direct contacts with the clinical staff. Follow up study finished in 2008.
Sampling Method: Non-Probability Sample
Enrollment: 2342 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jozefiak, M.D., Principal Investigator — NTNU Norwegian University of Science and Technology
Locations (1):
- NTNU Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jozefiak T, Sonnichsen Kayed N. Self- and proxy reports of quality of life among adolescents living in residential youth care compared to adolescents in the general population and mental health services. Health Qual Life Outcomes. 2015 Jul 22;13:104. doi: 10.1186/s12955-015-0280-y. PMID 26197764
- [Result] Jozefiak T, Larsson B, Wichstrom L, Wallander J, Mattejat F. Quality of Life as reported by children and parents: a comparison between students and child psychiatric outpatients. Health Qual Life Outcomes. 2010 Nov 22;8:136. doi: 10.1186/1477-7525-8-136. PMID 21092189